CLINICAL TRIAL: NCT00155155
Title: Analysis of HBV-Specific T Cell Responses and Regulatory T Cells in Patients With Chronic Hepatitis B Virus Infection
Brief Title: Studies of Immune Responses in Patients With Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701122; NSC 94-3112-B-002-030
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2008-11

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Taiwan is a hyperendemic area of hepatitis B virus (HBV) infection. Previous studies demonstrated vigorous T cell responses to HBV-encoded antigens developed in patients with self-limited acute hepatitis B. In contrast, weak or no T cell responses could be detected in chronic hepatitis B (CH-B) patients. However, these immune responses are still not well known in patients with acute exacerbation (AE) of CH-B and in patients with advanced liver diseases, such as liver cirrhosis (LC) and hepatocellular carcinoma (HCC). The CD4+CD25+ regulatory T cells might suppress immune responses against foreign antigens and pathogens. The roles of CD4+CD25+ regulatory T cells in patients chronically infected with HBV remain to be clarified. The high percentage of HBV carriers in Taiwan are related to the vertical transmissions. High maternal HBV viral load may make the newborns tolerant to the HBV. However, the HBV-specific CD8+ T cells responses in the cord bloods of newborns are still unknown. Thus, we want to resolve these issues in this study. We will enroll the HBsAg (+) patients from NTUH. Blood samples will be collected. We will then analyze the HBV-specific CD8+ T cell responses and the clarify the roles of regulatory T cells.

DETAILED DESCRIPTION:
The HBsAg (+) patients from National Taiwan University Hospital will be included. Screening for HLA haplotype will be performed by amplification refractory mutation system / PCR method. The HLA-A2 or HLA-A11 will be enrolled to the study group because these two haplotypes are the most ones in Taiwan. The other HLA haplotype HBV carriers will be enrolled as HLA-mismatch control. The disease spectra include inactive HBV carrier, CH-B, CH-B with AE (defined as ALT >= 5 X UNL), HBV-related LC, HBV-related HCCs.

HBsAg, anti-HBs, IgM anti-HBc, HBeAg, anti-HBe, anti-HCV, anti-HDV, anti-HIV will be determined by commercial enzyme immunoassay kits. The serum levels of HBV DNA and genotypes will be done by quantitative real-time PCR. Patients who are also infected with HDV or HCV or HIV will be excluded.

PBMCs will be isolated from heparinized blood samples by density gradient centrifugation on Ficoll-Hypaque. The PBMC will be washed with phosphate-buffered saline (PBS) and resuspended in T cell medium.

Analysis of HBV-specific CD8+ T cell responses will be done by flow cytometry using pentamer staining.

To analyze HBV-specific CD8+ T cells responses in patients with chronic HBV infection (prospective study). This part of the study is to clarify the role of HBV-specific T cell responses during the course of acute exacerbation of CH-B. Blood will be collected at four important time points.

ELIGIBILITY:
Inclusion Criteria:

* patients chronically infected with hepatitis B virus

Exclusion Criteria:

* coinfected with HCV or HIV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan